CLINICAL TRIAL: NCT00846170
Title: Double Blind Placebo Controlled Study of the Effect of Probiotics "Co-Biotic" (TM)on Symptoms and Fecal Bacterial Composition in IBS Patients
Brief Title: Probiotics in Irritable Bowel Syndrome
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: sponsor decided they are not interested in the study due to finacial reasons
Sponsor: Meir Medical Center (Other)
Responsible Party: Professor Fred Konokoff, Meir Medical center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PB-01-09
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2011-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- probiotics (Active Comparator): patients with IBS that will receive investigational treatment for 4 weeks
  Interventions: Drug: co-biotic
- Placebo (Placebo Comparator): cross over of patients from arm 1
  Interventions: Drug: placebo 2T/day

INTERVENTIONS:
Drug: co-biotic — give probiotic 2 t/day
  Arms: probiotics
Drug: placebo 2T/day — cross over of patients from study arm to placebo arm
  Arms: Placebo

SUMMARY:
Probiotics are defined as 'mono- or mixed cultures of live micro-organisms which, when applied to animal or man, beneficially affect the host by improving the properties of the indigenous flora'. Certain probiotics possess potent antibacterial and antiviral properties. Probiotic antibacterial activity may derive from the direct secretion of bacteriocins, the elaboration of proteases directed against bacterial toxins or through their ability to adhere to epithelial cells and thus exclude pathogens. The antiviral properties of some probiotic organisms, including the stimulation of interferon production, together with the well-documented efficacy of certain probiotics in the therapy of rotavirus diarrhea suggests the potential for a role for these agents in PI-IBS. The efficacy of some probiotics in preferentially relieving 'gas-related' symptoms may be related to qualitative changes in the colonic flora, as described earlier, or through the suppression of Small intestinal bacterial overgrowth (SIBO) , as there are reports of efficacy of probiotics in SIBO.

The aim of the proposed study is to investigate whether the probiotic preparation "co biotic" can change the composition of fecal bile acids, fatty acids and bacterial composition, and whether such changes, if they occur, are correlated to a change in the symptoms of patients with IBS.

Materials and methods:

Patients diagnosed as having IBS by the Rome III criteria will be included in the study.

Study subjects will be interviewed by a physician who will asses the diagnosis of IBS according to the Rome III criteria. Subjects will sign an informed consent and fill an IBS questionnaire and a health related quality of life questionnaire,

A fecal sample will be obtained

The subject will receive the probiotic product in a dose of 2 tablets/day, or a placebo containing all the active ingredients in the probiotic capsule, besides the bacteria, for 4 weeks. They will then enter a washout period of 2 weeks in which they will not receive anything, and then another 4 weeks in which they will receive the probiotic product in a dose of 2 tablets/day, or a placebo. Patients will be randomized so that they will receive the study drug for 4 weeks and the placebo for 4 weeks, in a double-blinded fashion. Thus each patient will be his own control.

ELIGIBILITY:
Inclusion Criteria:

* IBS by Rome III criteria

Exclusion Criteria:

* other GI disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
clinical improvement as judged by IBS questionnaire, change in fecal bacterial composition secondary: change the composition of fecal bile acids, fatty acids and bacterial composition | 2 years
change the composition of fecal bile acids, fatty acids and bacterial composition | 1 year

SECONDARY OUTCOMES:
clinical improvement | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical center, Kfar Saba, Israel